CLINICAL TRIAL: NCT05031468
Title: Observational, Prospective Cohort Study of the Immunogenicity and Safety of SARS-CoV-2 Vaccines Administered During Pregnancy or Postpartum and Evaluation of Antibody Transfer and Durability in Infants
Brief Title: Multisite Observational Maternal and Infant Study for COVID-19
Acronym: MOMI-Vax
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Flor Munoz, Associate Professor, Baylor College of Medicine
Other Study IDs: STUDY00002767; 3UM1AI148576-02S5 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: COVID-19
Keywords: Immunization; Pregnancy; Lactation
MeSH Terms: conditions — COVID-19; Breast Feeding | interventions — Licensure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and breast milk samples will be collected from pregnant participants. Cord blood and serum samples will be collected from infant participants. Residual samples will be retained, for participants who consent to have these left over specimens used for secondary research studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1: Individuals vaccinated during pregnancy: Individuals who receive a Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) vaccine during pregnancy (up to 200 individuals per vaccine type)
  Interventions: Biological: Licensed or EUA SARS-CoV-2 vaccine
- Group 2: Individuals vaccinated postpartum: Individuals who receive a SARS-CoV-2 vaccine postpartum (up to 65 individuals per vaccine type)
  Interventions: Biological: Licensed or EUA SARS-CoV-2 vaccine
- Group 3: Infants of individuals vaccinated during pregnancy: Infants of individuals who receive a SARS-CoV-2 vaccine during pregnancy (approximately 200 infants per vaccine type)
  Interventions: Biological: Licensed or EUA SARS-CoV-2 vaccine
- Group 4: Infants of individuals vaccinated postpartum: Infants of individuals who receive a SARS-CoV-2 vaccine postpartum (approximately 65 infants per vaccine type)
  Interventions: Biological: Licensed or EUA SARS-CoV-2 vaccine
- Group 5: Individuals receiving additional vaccines during pregnancy: Individuals who receive additional SARS-CoV-2 vaccine(s), beyond the primary series, during pregnancy (up to 200 individuals).
  Interventions: Biological: Licensed or EUA SARS-CoV-2 vaccine
- Group 6: Infants of individuals receiving additional vaccines during pregnancy: Infants of individuals who received additional SARS-CoV-2 vaccine(s), beyond the primary series, during pregnancy (approximately 200 infants).
  Interventions: Biological: Licensed or EUA SARS-CoV-2 vaccine

INTERVENTIONS:
Biological: Licensed or EUA SARS-CoV-2 vaccine — Several SARS-CoV-2 vaccines utilizing different platforms (e.g., mRNA, viral vector, etc.), are available under EUA (and soon to be licensed) and are being administered to individuals who are pregnant or postpartum who belong to high-risk priority groups for vaccination. Participants will receive the SARS-CoV-2 vaccine of their choice or the type that is available to them. The researchers anticipate including up to 3 vaccines, whether given as part of the primary series or additional doses, as part of this non-interventional study.

SUMMARY:
This is an observational, non-interventional, prospective cohort study designed to collect clinical information and specimens to evaluate the immune responses from pregnant individuals and postpartum individuals and their infants following maternal receipt of licensed or Emergency Use Authorization (EUA) severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccines.

DETAILED DESCRIPTION:
SARS-CoV-2, the novel coronavirus that causes Coronavirus Disease 2019 (COVID-19) disease, first emerged in Wuhan, China in December 2019 and has continued to spread globally. SARS-CoV-2 is highly transmissible between humans. A number of public health measures, including social distancing, avoidance of large congregations, particularly indoors, and the wearing of face masks, have been introduced to prevent spread of the virus. However, once these measures are relaxed, unless population immunity exceeds herd immunity thresholds, recrudescence of SARS-CoV-2 is expected. This underscores the urgent need for a safe and effective SARS-CoV-2 vaccine.

While all vaccines in late-stage development are based on the SARS-CoV- 2 S glycoprotein, they differ in other important characteristics, including manufacturing platform, number of doses, and immunogenicity and safety profiles. Two messenger RNA (mRNA)-based vaccines BNT162b2 (Pfizer-BioNTech) and mRNA-1273 (NIAID-Moderna) were granted Emergency Use Authorization (EUA) by the U.S. FDA based on high demonstrated efficacy against symptomatic infection and severe disease in diverse populations. Janssen (Johnson & Johnson) was also granted EUA for their single dose nonreplicating adenovirus vector vaccine. None of these large vaccine trials enrolled pregnant or lactating women (except for a small number of lactating women who were enrolled in the Janssen study).

The mRNA vaccines are being distributed to prioritized population groups, and other vaccines are expected to follow as they receive EUA approval. The Centers for Disease Control and Prevention (CDC) Advisory Committee on Immunization Practices (ACIP) gave a permissive recommendation for pregnant individuals who are in a priority group to receive SARS-CoV-2 vaccines based on risk of exposure or comorbidities. In addition, some states have included pregnant individuals in priority groups based on pregnancy itself being considered a high-risk condition by CDC. Thus, pregnant individuals are choosing to receive these vaccines under EUA, without trial data on safety and efficacy. There are neither data on the safety of SARS-CoV-2 vaccines in lactating women nor on the effects of mRNA or other vaccines on the breastfed infant or on milk production/excretion. Current EUA vaccines are not thought to be a risk to the breastfeeding infant.

Currently, additional doses of SARS-CoV-2 vaccines are being considered to enhance durability and breadth of protection, particularly against variant strains. On August 25, 2021, Pfizer submitted a supplement to their Biologics License Application (BLA) for their mRNA vaccine seeking approval for administration of an additional dose, and other manufacturers are expected to follow. In the setting of this rapidly evolving regulatory and policy environment, it is important that data on kinetics and durability of maternal and infant antibodies be generated for all vaccine regimens, including any additional doses beyond the primary series that may be administered to pregnant women.

Vaccines for pregnant individuals, such as influenza, tetanus and pertussis vaccines, are one of the most important public health measures globally to reduce disease in both mothers and infants in the first months of life. Various organizations support the position that pregnant and lactating women are a priority population and must not be excluded from the SARS-CoV-2 vaccine allocation strategy.

The purpose of this study is to evaluate the immunogenicity and safety of various licensed or EUA SARS-CoV-2 vaccines administered to pregnant or lactating women and describe the transplacental antibody transfer and kinetics of antibodies in infants. The researchers will also evaluate the durability of the antibodies in mothers and infants and assess breast milk antibodies in lactating women. The researchers will evaluate breast milk antibodies to assess potential for protection against COVID-19 in breastfed infants, similar to influenza vaccine protection from influenza illness in infants of mothers vaccinated during pregnancy or postpartum. The researchers anticipate including up to 3 vaccines, whether given as part of the primary series or additional doses, as part of this non-interventional study. It is expected that the results of this study will inform policy recommendations and personal decision-making on the use of approved SARS-CoV-2 vaccines in pregnant and lactating individuals.

This is an observational, non-interventional, prospective cohort study designed to collect clinical information and specimens to evaluate the immune responses from approximately 2,000 study participants following maternal receipt of licensed or EUA SARS-CoV-2 vaccines. Participants receiving a SARS-CoV-2 vaccine either during pregnancy or within 2 months of delivery, and their infants, will be followed for 12 months after delivery.

ELIGIBILITY:
Inclusion Criteria for Pregnancy Group (Group 1):

* Pregnant individuals who are scheduled to receive or have received complete vaccination series of any licensed or EUA SARS-CoV-2 vaccine during pregnancy. (NOTE: no limitation health status, or gestational age at enrollment)
* Willing and able to provide consent for study participation for herself and for her infant prior to initiation of any study procedures.

Inclusion Criteria for Postpartum Group (Group 3):

* Individuals who are scheduled to receive or who have initiated vaccination series of any licensed or EUA SARS-CoV-2 vaccine within the first 2 months postpartum. (NOTE: no limitation on health status).
* Willing and able to provide consent for study participation for herself and for her infant prior to initiation of any study procedures (a separate consent form will be used for their infants).

Inclusion Criteria for Additional Dose(s) During Pregnancy Group (Group 5):

* Pregnant individuals who received one dose or both doses of their primary vaccine series prior to pregnancy and are scheduled to receive or have received additional dose(s) of any licensed or EUA SARS-CoV-2 vaccine during pregnancy OR pregnant individuals who received complete vaccination series during pregnancy and are scheduled to receive or have received additional dose(s) of any licensed or EUA SARS-CoV-2 vaccine during pregnancy. (NOTE: no limitation on health status or gestational age at enrollment). This applies to individuals who have completed their primary series and receive an additional dose during pregnancy.
* Willing and able to provide consent for study participation for herself and for her infant prior to initiation of any study procedures.

Inclusion Criteria for All Participants:

* ≥18 years of age at time of enrollment
* Understands and agrees to comply with all study procedures.
* Agrees to sign medical release for herself and her infant to allow study staff to gather pertinent medical information, pregnancy outcome data, and medical information as needed.

Exclusion Criteria:

* Behavioral (including a history of alcohol or drug abuse within 1 year prior to study enrollment) or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
* Any condition which, in the opinion of the investigators, may pose a health risk to the subject or interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant individuals and postpartum individuals (within 2 months of delivery) who will be or have been vaccinated with a licensed or EUA SARS-CoV-2 vaccine, and their infants will be enrolled. Individuals receiving additional SARS-CoV-2 vaccine (beyond the primary series) during pregnancy will also be enrolled. Upon delivery, the infants born to individuals who received vaccine during pregnancy will become study participants.
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Change in Geometric Mean Titer (GMT) of Serum Immunoglobulin G (IgG) Among Individuals Vaccinated During Pregnancy | Baseline, 28 days post-vaccination, at delivery, postpartum months 2, 6, and 12
  The kinetics and durability of maternal serum antibodies following receipt of SARS-CoV-2 vaccine during pregnancy will be assessed as the GMT of IgG enzyme-linked immunosorbent assay (ELISA), by vaccine type and/or platform (mRNA, viral vector, etc.).
Change in GMT of Neutralizing (Neut) Antibodies in Serum Among Individuals Vaccinated During Pregnancy | Baseline, 28 days post-vaccination, at delivery, postpartum months 2, 6, and 12
  The kinetics and durability of maternal serum antibodies following receipt of SARS-CoV-2 vaccine during pregnancy will be assessed as the GMT of Neut antibodies by vaccine type, platform and dose regimen.
GMT of Cord Blood IgG | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the GMT of IgG in cord blood, overall and by vaccine type, platform and dose regimen.
Ratio of Cord Blood IgG to Maternal Serum IgG | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the ratio of cord blood IgG to maternal serum IgG, overall and by vaccine type, platform and dose regimen.
Neut antibodies of cord blood | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the GMT of Neut antibodies in cord blood, overall and by vaccine type, platform and dose regimen.
Ratio of cord blood Neut antibodies to maternal serum Neut antibodies | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the ratio of cord blood Neut antibodies to maternal Neut antibodies, overall and by vaccine type and platform.
Change GMT of serum IgG in Infants Born to Individuals Vaccinated During Pregnancy | At delivery, 2 months of age, 6 months of age
  The kinetics and durability of serum SARS-CoV-2 antibodies in infants of mothers vaccinated during pregnancy will be assessed as the GMT of IgG in infants, by vaccine type, platform and dose regimen.
Change GMT of Neut antibodies in Infants Born to Individuals Vaccinated During Pregnancy | At delivery, 2 months of age, 6 months of age
  The kinetics and durability of serum SARS-CoV-2 antibodies in infants of mothers vaccinated during pregnancy will be assessed as the GMT of Neut antibodies in infants, by vaccine type, platform and dose regimen.

SECONDARY OUTCOMES:
Frequency of Maternal Outcomes | At delivery
  The frequency of maternal outcomes among individuals receiving the SARS-CoV-2 vaccine during pregnancy or postpartum will be compared to background rates in the United States, overall and by vaccine type and platform.
Frequency of Infant Outcomes | At delivery
  The frequency of infant outcomes among infants born to individuals receiving the SARS-CoV-2 vaccine during pregnancy or postpartum will be compared to background rates in the United States, overall and by vaccine type and platform.
GMT of Serum IgG Compared to Non-Pregnant Women | 28 days post-vaccination
  GMT of Serum IgG in individuals receiving different SARS-CoV-2 vaccines during pregnancy or postpartum will be compared to non-pregnant populations of women of childbearing age.
GMT of Neut Antibodies Compared to Non-Pregnant Women | 28 days post-vaccination
  GMT of Neut antibodies in individuals receiving different SARS-CoV-2 vaccines during pregnancy or postpartum will be compared to non-pregnant populations of women of childbearing age.
GMT of Serum IgG by Gestational Age at Vaccination | 28 days post-vaccination
  GMT of serum IgG in individuals receiving different SARS-CoV-2 vaccines during pregnancy will be examined by gestational age at vaccination (trimester of gestation) and interval between vaccination and delivery, by vaccine type and platform.
GMT of Neut Antibodies by Gestational Age at Vaccination | 28 days post-vaccination
  GMT of Neut antibodies in individuals receiving different SARS-CoV-2 vaccines during pregnancy will be examined by gestational age at vaccination (trimester of gestation) and interval between vaccination and delivery, by vaccine type and platform.
GMT of Serum IgG by Baseline Characteristics | 28 days post-vaccination
  GMT of serum IgG in individuals receiving different SARS-CoV-2 vaccines during pregnancy or postpartum will be examined by maternal age, health status, and risk status (e.g., occupation, priority vaccination group) overall and by vaccine type and platform.
GMT of Neut Antibodies by Baseline Characteristics | 28 days post-vaccination
  GMT of Neut antibodies in individuals receiving different SARS-CoV-2 vaccines during pregnancy or postpartum will be examined by maternal age, health status, and risk status (e.g., occupation, priority vaccination group) overall and by vaccine type and platform.
GMT of Cord Blood IgG by Gestational Age at Vaccination | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the GMT of IgG in cord blood, by gestational age at vaccination (trimester of vaccination) and interval between vaccination and delivery, overall and by vaccine type and/or platform.
Ratio of Cord Blood IgG to Maternal Serum IgG by Gestational Age at Vaccination | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the ratio of cord blood IgG to maternal serum IgG, by gestational age at vaccination (trimester of vaccination) and interval between vaccination and delivery, overall and by vaccine type and/or platform.
GMT of Cord Blood Neut Antibodies by Gestational Age at Vaccination | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the GMT Neut antibodies in cord blood, by gestational age at vaccination (trimester of vaccination) and interval between vaccination and delivery, overall and by vaccine type and/or platform.
Ratio of Cord Blood Neut Antibodies to Maternal Serum Neut Antibodies by Gestational Age at Vaccination | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the ratio of cord blood Neut antibodies to maternal Neut antibodies, by gestational age at vaccination (trimester of vaccination) and interval between vaccination and delivery, overall and by vaccine type and/or platform.
GMT of Cord Blood IgG by Baseline Characteristics | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the GMT of IgG in cord blood, by maternal age, health status, and risk status (e.g., occupation, priority vaccination group) overall and by vaccine type and platform.
Ratio of Cord Blood IgG to Maternal Serum IgG by Baseline Characteristics | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the ratio of cord blood IgG to maternal serum IgG, by maternal age, health status, and risk status (e.g., occupation, priority vaccination group) overall and by vaccine type and platform.
GMT of Cord Blood Neut Antibodies by Baseline Characteristics | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the GMT Neut antibodies in cord blood, by maternal age, health status, and risk status (e.g., occupation, priority vaccination group) overall and by vaccine type and platform.
Ratio of Cord Blood Neut Antibodies to Maternal Serum Neut Antibodies by Baseline Characteristics | At delivery
  Transplacental antibody transfer of SARS-CoV-2 antibodies among individuals vaccinated during pregnancy will be assessed as the ratio of cord blood Neut antibodies to maternal Neut antibodies, by maternal age, health status, and risk status (e.g., occupation, priority vaccination group) overall and by vaccine type and platform.
Change in GMT of IgG in Breast Milk | 2 weeks postpartum, and 2, 6, and 12 months postpartum
  The kinetics of SARS-CoV-2 antibodies in breast milk of mothers who received vaccine during pregnancy or postpartum, will be assessed as the GMT of IgG in breast milk, overall and by vaccine type and platform.
Change in GMT of Immunoglobulin A (IgA) in Breast Milk | 2 weeks postpartum, and 2, 6, and 12 months postpartum
  The kinetics of SARS-CoV-2 antibodies in breast milk of mothers who received vaccine during pregnancy or postpartum, will be assessed as the GMT of IgA in breast milk, overall and by vaccine type and platform.
Change in GMT of Neut Antibodies in Breast Milk | 2 weeks postpartum, and 2, 6, and 12 months postpartum
  The kinetics of SARS-CoV-2 antibodies in breast milk of mothers who received vaccine during pregnancy or postpartum, will be assessed as the GMT of Neut Antibodies in breast milk, overall and by vaccine type and platform.
Change in GMT of Serum IgG Among Individuals Vaccinated Postpartum | Baseline, 28 days post-vaccination, postpartum months 2, 6, and 12
  The kinetics and durability of maternal serum antibodies following receipt of SARS-CoV-2 vaccine postpartum will be assessed as the GMT of IgG, by vaccine type and/or platform.
Change in GMT of Neutralizing (Neut) Antibodies in Serum Among Individuals Vaccinated Postpartum | Baseline, 28 days post-vaccination, postpartum months 2, 6, and 12
  The kinetics and durability of maternal serum antibodies following receipt of SARS-CoV-2 vaccine postpartum will be assessed as the GMT of Neut antibodies, by vaccine type and/or platform.
Change GMT of serum IgG in Infants Born to Individuals Vaccinated Postpartum | 2 months of age, 6 months of age
  The kinetics and durability of serum SARS-CoV-2 antibodies in infants of mothers vaccinated postpartum will be assessed as the GMT of IgG in infants, by vaccine type and platform.
Change GMT of Neut antibodies in Infants Born to Individuals Vaccinated Postpartum | 2 months of age, 6 months of age
  The kinetics and durability of serum SARS-CoV-2 antibodies in infants of mothers vaccinated postpartum will be assessed as the GMT of Neut antibodies in infants, by vaccine type and platform.
Change in GMT of Serum IgG Among Individuals Receiving Additional Vaccine Dose(s) | Baseline, 28 days post-vaccination, postpartum months 2, 6, and 12
  The kinetics and durability of maternal serum antibodies following receipt of additional dose(s) of SARS-CoV-2 vaccine in pregnant individuals who received vaccine prior to pregnancy, will be assessed as the GMT of IgG in serum, by vaccine type and platform.
Change in GMT of Neut Antibodies Among Individuals Receiving Additional Vaccine Dose(s) | Baseline, 28 days post-vaccination, postpartum months 2, 6, and 12
  The kinetics and durability of maternal serum antibodies following receipt of additional dose(s) of SARS-CoV-2 vaccine in pregnant individuals who received vaccine prior to pregnancy, will be assessed as the GMT of Neut antibodies, by vaccine type and platform.

OTHER OUTCOMES:
Incidence of COVID-19 Infection Among Pregnant Individuals | Up to postpartum month 12
  The effectiveness of SARS-CoV-2 vaccines against maternal COVID-19 infection during pregnancy and postpartum will be assessed as the incidence of laboratory confirmed COVID-19 illness during study participation assessed through passive surveillance in individuals vaccinated during pregnancy or postpartum compared to rates in unvaccinated women of childbearing age, overall and by vaccine type and platform.
Severity of COVID-19 Infection Among Pregnant Individuals | Up to postpartum month 12
  The effectiveness of SARS-CoV-2 vaccines against maternal COVID-19 infection during pregnancy and postpartum will be assessed as the severity of COVID-19 disease during study participation assessed through passive surveillance in individuals vaccinated during pregnancy or postpartum compared to rates in unvaccinated women of childbearing age, overall and by vaccine type and platform.
Incidence of COVID-19 Infection Among Infants | Up to 12 months of age
  The effectiveness of maternal antibodies to provide protection against SARS-CoV-2 will be assessed by examining the incidence of COVID-19 illness in infants in the first 12 months of life. Incidence of laboratory confirmed COVID-19 during study participation is assessed through passive surveillance in infants of individuals vaccinated in pregnancy or postpartum compared to background rates in infants of unvaccinated women of childbearing age, overall and by vaccine type and platform.
Severity of COVID-19 Infection Among Infants | Up to 12 months of age
  The effectiveness of maternal antibodies to provide protection against SARS-CoV-2 will be assessed by examining the severity of COVID-19 illness in infants in the first 12 months of life. The severity of laboratory confirmed COVID-19 during study participation is assessed through passive surveillance in infants of individuals vaccinated in pregnancy or postpartum vs. background rates in infants of unvaccinated women of childbearing age, overall and by vaccine type and platform.
Incidence of COVID-19 Infection Among Breastfed Infants | Up to 12 months of age
  The effectiveness of breastmilk antibodies to provide protection against SARS-CoV-2 will be assessed by examining the incidence of COVID-19 illness in infants in the first 12 months of life. The incidence of laboratory confirmed COVID-19 during study participation is assessed through passive surveillance in breastfed infants compared to not breastfed infants, by vaccine type and platform.
Severity of COVID-19 Infection Among Breastfed Infants | Up to 12 months of age
  The effectiveness of breastmilk antibodies to provide protection against SARS-CoV-2 will be assessed by examining the severity of COVID-19 illness in infants in the first 12 months of life. The severity of laboratory confirmed COVID-19 during study participation is assessed through passive surveillance in breastfed infants compared to not breastfed infants, by vaccine type and platform.
Incidence of COVID-19 Infection Among Breastfed Infants by Vaccination Timing | Up to 12 months of age
  The effectiveness of breastmilk antibodies to provide protection against SARS-CoV-2 will be assessed by examining the severity of COVID-19 illness in infants in the first 12 months of life. The severity of laboratory confirmed COVID-19 during study participation is assessed through passive surveillance in breastfed infants of individuals vaccinated during pregnancy compared to postpartum, overall and by vaccine type and platform.
Severity of COVID-19 Infection Among Breastfed Infants by Vaccination Timing | Up to 12 months of age
  The effectiveness of breastmilk antibodies to provide protection against SARS-CoV-2 will be assessed by examining the severity of COVID-19 illness in infants in the first 12 months of life. The severity of laboratory confirmed COVID-19 during study participation is assessed through passive surveillance in breastfed infants of individuals vaccinated during pregnancy compared to postpartum, overall and by vaccine type and platform.

CONTACTS AND LOCATIONS:
Overall Officials: Flor Munoz, MD, Principal Investigator — Baylor College of Medicine
Locations (10):
- United States (10):
  - Emory University, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - New York University Langone Vaccine Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Magee - Womens Hospital, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available for sharing for secondary research, following de-identification.
Supporting Information: SAP, Analytic Code
Time Frame: Data will be available for sharing immediately following publication of the results of this study, with no end date, with data sharing at the discretion of the Infectious Diseases Clinical Research Consortium (IDCRC).
Access Criteria: Data will be made available for sharing for secondary research with investigators/researchers upon written request, with provision of a methodologically sound proposal. The proposal will need approval from Division of Microbiology and Infectious Diseases (DMID) and any approvals required by the site or consortium. The data will be available for only the purpose outlined in the approved proposal. Proposals can be sent to Dr. Munoz at florm@bcm.edu.

REFERENCES:
- [Background] Munoz FM, Beigi RH, Posavad CM, Richardson BA, Chu HY, Bok K, Campbell J, Cardemil C, DeFranco E, Frenck RW, Makhene M, Piper JM, Sheffield J, Miller A, Neuzil KM. Multi-site observational maternal and infant COVID-19 vaccine study (MOMI-vax): a study protocol. BMC Pregnancy Childbirth. 2022 May 12;22(1):402. doi: 10.1186/s12884-022-04500-w. PMID 35550037
- [Result] Munoz FM, Posavad CM, Richardson BA, Badell ML, Bunge K, Mulligan MJ, Parameswaran L, Kelly C, Olsen-Chen C, Novak RM, Brady RC, Pasetti M, DeFranco E, Gerber JS, Shriver M, Suthar MS, Moore K, Coler R, Berube B, Kim SH, Piper JM, Miller A, Cardemil C, Neuzil KM, Beigi R; DMID Study Group. COVID-19 booster vaccination during pregnancy enhances maternal binding and neutralizing antibody responses and transplacental antibody transfer to the newborn (DMID 21-0004). medRxiv [Preprint]. 2022 Jun 13:2022.06.13.22276354. doi: 10.1101/2022.06.13.22276354. PMID 35734087
- [Result] Cardemil CV, Cao Y, Posavad CM, Badell ML, Bunge K, Mulligan MJ, Parameswaran L, Olson-Chen C, Novak RM, Brady RC, DeFranco E, Gerber JS, Pasetti M, Shriver M, Coler R, Berube B, Suthar MS, Moreno A, Gao F, Richardson BA, Beigi R, Brown E, Neuzil KM, Munoz FM; MOMI-Vax Study Group. Maternal COVID-19 Vaccination and Prevention of Symptomatic Infection in Infants. Pediatrics. 2024 Mar 1;153(3):e2023064252. doi: 10.1542/peds.2023-064252. PMID 38332733